CLINICAL TRIAL: NCT00306059
Title: Early Goal Directed Therapy for Acute Kidney Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigators decision
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006/096
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Kidney Injury, Acute
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients having acute kidney injury (Experimental)
  Interventions: Procedure: Early goal directed therapy during 6 hours after occurence of the early phase of acute kidney injury

INTERVENTIONS:
Procedure: Early goal directed therapy during 6 hours after occurence of the early phase of acute kidney injury — Directed therapy during 6 hours after occurence of the early phase of acute kidney injury.

SUMMARY:
Early goal directed therapy during 6 hours after occurence of the early phase of acute kidney injury

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* occurence of the early phase of acute kidney injury
* stay on intensive care unit

Exclusion Criteria:

* chronic haemodialysis
* not given informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Observation of acute kidney injury | after 48 hours

SECONDARY OUTCOMES:
Organ failure during first 48 hours and during stay on intensive care unit | after 48 hours
Duration of stay on intensive care unit and in hospital | t0
Mortality during stay on intensive care unit | after 28 days, 60 days and during stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hoste, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be